CLINICAL TRIAL: NCT01979796
Title: Antismoking Effects of Electronic Cigarettes in Subjects With Schizophrenia and Their Potential Influence on Cognitive Functioning: Design of a Randomized Trial. Smoking Cessation And Reduction In Schizophrenia (The SCARIS Study)
Brief Title: Antismoking Effects of Electronic Cigarettes in Subjects With Schizophrenia and Their Potential Influence on Cognitive Functioning.
Acronym: SCARIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universita degli Studi di Catania (Other)
Responsible Party: Principal Investigator, Riccardo Polosa, Professor, Universita degli Studi di Catania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCARIS
Record Dates: First submitted 2013-10-24; First posted 2013-11-08 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Tobacco Smoking in Schizophrenic Patients
Keywords: Addiction, Schizophrenia, Electronic cigarettes
MeSH Terms: conditions — Behavior, Addictive; Schizophrenia; Vaping | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ecig 24 mg nicotine (Experimental): Ecig 24 mg nicotine
  Interventions: Device: Ecig 24 mg nicotine
- Ecig 0 mg nicotine (Sham Comparator): Ecig 0 mg nicotine
  Interventions: Device: Ecig 0 mg nicotine
- Nicotine free inhalator (Placebo Comparator): Nicotine free inhalator
  Interventions: Device: Nicotine free inhalator

INTERVENTIONS:
Device: Ecig 24 mg nicotine — Cigalike
  Arms: Ecig 24 mg nicotine
Device: Ecig 0 mg nicotine — Cigalike
  Arms: Ecig 0 mg nicotine
Device: Nicotine free inhalator — Plastic CIG a Like
  Arms: Nicotine free inhalator

SUMMARY:
It is well established in studies across several countries that tobacco smoking is more prevalent among schizophrenic patients than the general population. Electronic cigarettes (e-cigarettes) are becoming increasingly popular with smokers worldwide. To date there are no large randomised trials of e-cigarettes in schizophrenic smokers. A well-designed trial is needed to compare efficacy and safety of these products in this special population.

DETAILED DESCRIPTION:
The investigators have designed a randomized controlled trial investigating the efficacy and safety of electronic cigarette. The trial will take the form of a prospective 12-month randomized clinical study to evaluate smoking reduction, smoking abstinence and adverse events in schizophrenic smokers not intending to quit. The investigators will also monitor quality of life, neurocognitive functioning and measure participants' perception and satisfaction of the product.

The main strengths of the SCARIS study are the following: it's the first large RCT on schizophrenic patient, involving in and outpatient, evaluating the effect of a three-arm study design, and a long term of follow-up (52-weeks).

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenic subjects (according to DSM-IV-TR criteria) from throughout Sicily, (Italy), who smoke tobacco cigarettes, in stable phase of illness.
* smoke ≥10 factory made cig/day, for at least the past five years
* age 18-65 years
* in good general health
* not currently attempting to quit smoking or wishing to do so in the next 30 days (a specific test will be included to check their unwillingness to quit) 6 months
* committed to follow the trial procedures.

Exclusion Criteria:

* use of smokeless tobacco or nicotine replacement therapy
* pregnancy or breastfeeding.
* current or recent (less than 1 yr) past history of alcohol and/or drug abuse
* other significant co-morbidities according to the Investigator's clinical assessment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
smoking cessation | 52 weeks
  Abstinence from smoking, defined as complete self-reported abstinence from tobacco smoking - not even a puff (together with an eCO concentration of ≤7 ppm), will be calculated at each study visit ("quitters").

SECONDARY OUTCOMES:
Smoking reduction | 52 weeks
  A ≥50% reduction in the number of cig/day from baseline, defined as self-reported reduction in the number of cig/day (≥50%) compared to baseline (together with an eCO levels reduction, to objectively document a reduction from baseline), will be calculated at each study visit ("reducers").
  Smokers who will not satisfy the criteria of "reducers" and "quitters" will be defined "non responders".

OTHER OUTCOMES:
Evaluation of neurocognitive functioning | 52 weeks
  Quality of life, Neurocognitive Functioning and Psychopathological status will be assessed at each study visit by Quality of Life Scale (QLS), Brief Assessment of Cognition in Schizophrenia (BACS) and Positive and Negative Symptoms Scale(PANSS), respectively
  Participants' perception and liking of the product will be assessed by asking to rate their level of satisfaction with the products compared to their own cigarettes using a visual analogue scale (VAS) from 0 to 10 points (0 = being 'completely unsatisfied', 10 being = 'fully satisfied'); using the same scale, they will also rate how much they miss their own brand (0 = being 'did not miss it at all', 10 being = 'missed too much') and whether they would recommend it to a friend/relative (0 = being 'not recommended at all', 10 being = 'absolutely recommended').

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Caponnetto, Assis Prof, Principal Investigator — University of Catania; Eugenio Aguglia, Professor, Principal Investigator — University of Catania; Giuseppe Minutolo, Assis prof, Principal Investigator — University of Catania

REFERENCES:
- [Derived] Caponnetto P, Polosa R, Auditore R, Minutolo G, Signorelli M, Maglia M, Alamo A, Palermo F, Aguglia E. Smoking cessation and reduction in schizophrenia (SCARIS) with e-cigarette: study protocol for a randomized control trial. Trials. 2014 Mar 22;15:88. doi: 10.1186/1745-6215-15-88. PMID 24655473